CLINICAL TRIAL: NCT05306392
Title: Evaluation of the Effectiveness of Induced Moderate Hypothermia in the Management of Patients With Severe ARDS Under Venovenous ECMO
Brief Title: Effects of Induced Moderate Hypothermia on ARDS Patients Under Venovenous ExtraCorporeal Membrane Oxygenation
Acronym: HypoLungECMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Klein Thomas, Principal investigator, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A00168-35
Record Dates: First submitted 2022-02-16; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-02

CONDITIONS: ARDS, Human; Extracorporeal Membrane Oxygenation Complication; Hypothermia
Keywords: Hypothermia; ECMO; Refractory hypoxemia
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypothermia; Hypoxia | interventions — Hypothermia, Induced

STUDY DESIGN:
Intervention Model Description: Monocentric controlled study, with randomization in two groups (induced hypothermia group and control group), at the Nancy Hospital - Intensive care Unit
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Hypothermia (Experimental): Patients with acute respiratory distress syndrome treated with venovenous ECMO to a strategy of moderate hypothermia during 48 hours (Temperature at 33°C≤ T°C ≤34°C) associated with usual care
  Interventions: Device: Moderate Hypothermia
- Control - Normothermia (Sham Comparator): Patients with acute respiratory distress syndrome treated with venovenous ECMO to a strategy of normothermia (36°C≤ T°C ≤37°C) associated with usual care
  Interventions: Device: Normothermia

INTERVENTIONS:
Device: Moderate Hypothermia — moderate hypothermia will be induced using the heat controller of the VV-ECMO circuit. Temperature will be maintained between 33°C≤ T°C ≤34°C during 48 hours followed by a progressive reheating (0.2±0.1°C/h) to reach 36 °C. Temperature at 36°C will be maintained during 48 hours after having reached 36 °C.
  Arms: Moderate Hypothermia
Device: Normothermia — Temperature at 36°C will be maintained during 48 hours after having reached 36 °C
  Arms: Control - Normothermia

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a lesional pulmonary edema that occurs as a result of direct or indirect lung injury. This condition accounts for 10-15% of ICU admissions and 20-25% of patients admitted require invasive ventilation. Its incidence has increased markedly with the Covid-19 epidemic. ARDS is defined as hypoxemia (Pa02/Fi02 < 300 mmHg) in ventilated patients without heart failure. Currently, the recommendations of the resuscitation societies advocate a management combining invasive ventilation, short duration curarization and prone sessions. In case of failure of these therapies, venovenous ExtraCorporeal Membrane Oxygenation (VV ECMO) is recommended in case of Pa02/Fi02 < 80 mmHg.

Nevertheless, approximately 40% of patients have refractory and persistent hypoxemia despite optimization of ECMO parameters and invasive ventilation. The refractory hypoxemia is defined as Pa02 < 55 mmHg and/or Sa02 < 90% and may be due to a recirculation phenomenon or a significant intra-pulmonary shunt. Currently, there is no official recommendation for the management of these patients, leading to the use of various unvalidated field practices. In addition, hospital mortality of the order of 60% is observed in these patients with high management costs.

Some data in the literature suggest that induced therapeutic hypothermia (HT) at 34°C for 48 hours could improve the prognosis of these patients by improving oxygenation. Nevertheless, the level of evidence of published studies remains low because they are either case reviews or studies whose methodology does not guarantee the absence of potential bias.

The research hypothesis is that HT at 34°C or 33°C for 48 hours is effective on refractory hypoxemia.

DETAILED DESCRIPTION:
The investigators propose a pilot study, monocentric, prospective, controlled, randomized, to apprehend in an objective and reliable way the effects of induced moderate hypothermia at 34°C, or at 33°C in case of persistence of a Sa02 lower than 90%, during 48 hours in patients under ECMO VV for ARDS. The objective of this study is to show the beneficial effect of the treatment on the patient's oxygenation and to understand the physiopathological mechanism of action at work through different parameters at different times. In parallel, the undesirable effects will be recorded and weighed against the positive effects of the treatment in order to understand the benefit/risk ratio of light HT. The effect on survival will also be evaluated as a secondary objective, not to demonstrate efficacy in this small pilot trial, but to determine the size of the effect that can be expected.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Intubated, ventilated patients with ARDS requiring VV ECMO
* Family member or trusted person who has been informed about the study and signed the informed consent form or inclusion in an immediate life-threatening situation
* Benefiting from a Social Security affiliation scheme

Exclusion Criteria:

* Presence of a recirculation phenomenon (distance between the 2 ECMO cannulas < 10 cm).
* Patients expected to die within 48 hours of VV ECMO implantation
* Patients on short-acting beta blockers
* Pregnant, parturient or lactating woman,
* Persons deprived of their liberty by a judicial or administrative decision,
* Minors (non emancipated)
* Adults subject to legal protection measures (guardianship, curatorship, safeguard of justice).
* Person undergoing psychiatric care under articles L3212-1 and L3213-1 of the french Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of 48 hours therapeutic hypothermia on the evolution of hypoxemia in patients on VV ECMO | between initiation of hypothermia and 48 hours of induced hypothermia
  Hypoxemia is measured by arterial saturation of oxygen (expressed in %)

SECONDARY OUTCOMES:
Effectiveness of 1 hours, 6 hours, 24 hours therapeutic hypothermia on the evolution of hypoxemia in patients on VV ECMO | at 1 hour, 6 hours, 24 hours of the randomization
  Hypoxemia is measured by arterial saturation of oxygen (expressed in %)
Evolution of arterial transport of oxygen during therapeutic hypothermia | Evaluation of arterial transport of oxygen by peripheral gas measurement at 1 hour, 6 hours, 24 hours and 48 hours of hypothermia
  Arterial transport of oxygen is measured by blood gas at different hours (expressed in mL · min-1 · m-2)
Evolution of ECMO flow / cardiac output ratio (expressed in %) | Measurement at 1 hour, 6 hours, 24 hours and 48 hours
  Evaluation of the impact of induced hypothermia on the evolution of the ratio of ECMO flow (expressed in L/min) to the patient's cardiac output (assessed by cardiac ultrasound and expressed in L/min).
  The ratio of ECMO output to patient's cardiac output (expressed in percentage) is calculated as the ratio of ECMO output (expressed in L/min) to cardiac output (expressed in L/min)
Survival of patients hospitalized in intensive care | Measurement following inclusion with a time maximal of 28 days
  The percentage of patients who died during resuscitation hospitalization
The duration of VV ECMO during hospitalization in the intensive care unit | Measurement following inclusion with a time maximal of 28 days
  The duration of VV ECMO (in days) during resuscitation hospitalization,
The number of days without mechanical ventilation during resuscitation hospitalization | Measurement following inclusion with a time maximal of 28 days
  The number of days without invasive mechanical ventilation during resuscitation hospitalization
Microcirculatory perfusion and flow variables | at 24 and 48 hours
  measurement of sublingual microcirculation by using Sidestream Dark Field (SDF) microscopy
  SDF will be applied to the sublingual microvascular network with a 5X objective providing a 167X magnification.
  After the removal of saliva and other secretions using gauze, the device will be gently applied (without any pressure) on the lateral side of the tongue, in an area approximately 1.5-4 cm from the tip of the tongue. Five sequences of 20 secs each from different adjacent areas will be recorded using a computer and a video card and stored under a random number for later analysis.
  Other Name: SDF ((Microscan; Microvision Medical, Amsterdam, the Netherlands)
The safety of induced hypothermia treatment during hospitalization in the intensive care unit (infections, coagulation disorders, cardiac risk). | Measurement following inclusion with a time maximal of 28 days
  For infectious risk: % of infections during hospitalization in the intensive care unit (maximum follow-up time of 28 days);
  For risk on coagulation:
  (i) plasma free hemoglobinemia (expressed in g per 100 mL), and on (ii) prothrombin level (expressed in %), at 48 hours; (iii) Need for blood transfusion with hemoglobin loss of more than 2 points within 48 hours of hypothermia (expressed in number of blood transfusion) (iv) Bleeding manifestations within 48 hours with or without need for surgical treatment;
  For cardiac risk:
  (i) percentage of patients with symptomatic cardiac rhythm disturbance requiring specific treatment between H0 and H24 and between H0 and H48 (expressed in percentage), (ii) total duration of vasopressors administered at H24 and at H48 (expressed in days)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno LEVY, PhD, Study Director — CHRU NANCY, Nancy, France; Nathalie THILLY, PhD, Study Chair — CHRU NANCY, Nancy, France; Thomas KLEIN, MD, Study Chair — CHRU NANCY, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Montisci A, Maj G, Zangrillo A, Winterton D, Pappalardo F. Management of refractory hypoxemia during venovenous extracorporeal membrane oxygenation for ARDS. ASAIO J. 2015 May-Jun;61(3):227-36. doi: 10.1097/MAT.0000000000000207. PMID 25923575
- [Result] Levy B, Taccone FS, Guarracino F. Recent developments in the management of persistent hypoxemia under veno-venous ECMO. Intensive Care Med. 2015 Mar;41(3):508-10. doi: 10.1007/s00134-014-3579-y. Epub 2014 Dec 2. No abstract available. PMID 25447805
- [Result] Kimmoun A, Vanhuyse F, Levy B. Improving blood oxygenation during venovenous ECMO for ARDS. Intensive Care Med. 2013 Jun;39(6):1161-2. doi: 10.1007/s00134-013-2903-2. Epub 2013 Apr 13. No abstract available. PMID 23584469